CLINICAL TRIAL: NCT03397433
Title: ANti-infective Stewardship Using the Wisca Tool in the Electronic Medical Record
Acronym: ANSWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EH13-368
Record Dates: First submitted 2017-12-29; First posted 2018-01-12 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Bacterial Infections
Keywords: Antibiotic Stewardship; Information Technology; Healthcare Outcomes; Antibiotic Resistance; Bacterial Infection
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Intervention Model Description: This is a prospective, pragmatic trial of initial antibiotic prescribing review by Infectious Disease Specialists. The study involves 4 hospitals, 2 of which are intervention and 2 control for 18 months, followed by switching the intervention and control hospitals in a crossover fashion for another 18 months. Medical and economic outcomes will be assessed and reported
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): In this arm, an Information Technology physician assist tool will be used to predict best available therapy for patients coming to the hospital with either pneumonia, cellulitis, intraabdominal infection, or complicated urinary tract infection.
  Intervention: After review of the information technology recommendation by a board certified Infectious Disease physician, the recommendation will be discussed with the primary care physician and treatment implemented.
  Interventions: Other: Information Technology physician assist
- Control (No Intervention): In the two control hospitals there will be no use of the information technology tool for implementation of initial treatment (No intervention). No notes will be placed in the electronic health record and no contact as a result of this research will be made with the medical care team.

INTERVENTIONS:
Other: Information Technology physician assist — The intervention hospitals will have a progress note placed in the electronic health record by a reviewing Infectious Disease specialist that comments on the initial antibiotic choice. The comment is based on an electronic prediction tool (Information Technology physician assist) as to what the best therapy is for the individual patient whose health record is reviewed.
  Arms: Intervention

SUMMARY:
Beginning in the mid-to late 1980s and accelerating through the 1990s and 2000s the shield of antibiotic invincibility began to crack sufficiently so that it was apparent to everyone we faced a serious problem. The investigators will demonstrate and expand the use of information technology based on the ingenious weighted-incidence, syndromic, combination antibiogram (WISCA) tool for the widespread use of automated clinician prompts enhancing empiric antibiotic therapy as part of a comprehensive infection control stewardship program that reduces antibiotic resistance. This research program will demonstrate that use of such a tool lowers mortality, improves outcome, lowers antimicrobial resistance and reduces healthcare cost.

DETAILED DESCRIPTION:
The decade of the 1970s was a time when the PI was completing his training and beginning a career in Infectious Diseases and Microbiology. This was an era when many new anti-infective compounds were being introduced, ranging from novel penicillins to extended-spectrum cephalosporins to aminoglycosides. The main antimicrobial resistance concern at the time was Staphylococcus aureus that was no longer susceptible to penicillin; methicillin, oxacillin, and nafcillin had solved that problem. Even for those strains that later were methicillin-resistant (MRSA), vancomycin had been available since the 1950s. Later the carbapenems and in the 1980s the newer fluoroquinolones, beginning with ciprofloxacin, were introduced for clinical use. At the time it seemed that the challenge of treating serious infection in humans had been met and that other diseases were a higher priority. Indeed, in 1978 one of the world's leaders in infectious diseases, Dr. Robert Petersdorf, commented that "Even with my great personal loyalty to Infectious Disease, I cannot conceive of the need for 309 more [graduating trainees in] infectious disease...unless they spend their time culturing each other". However, in Alexander Fleming's 1945 Nobel prize lecture he warned of the danger of antimicrobial resistance stating "it is not difficult to make microbes resistant to penicillin in the laboratory by exposing them to concentrations not sufficient to kill them, and the same thing has occurred occasionally happen in the body . . . and by exposing (his) microbes to nonlethal quantities of the drug make them resistant". It was also at this time that Infection Control began as an established discipline with CDC offering the first course in 1968 and the Joint Commission requiring a hospital position for Infection Control in 1969. Subsequently, beginning in the mid-to late 1980s and accelerating through the 1990s and 2000s the shield of antibiotic invincibility began to crack sufficiently so that it was apparent to everyone we faced a serious problem. Resistance began to be reported in Gram negative bacteria toward the newer cephalosporin, fluoroquinolone, and even the carbapenem drugs. During this same period modern medicine witnessed the emergence and spread of a new healthcare associated infection called Clostridium difficile associated diarrhea, as well as MRSA becoming pandemic. It was during this time that the initial studies focused on reversing antimicrobial resistance began. In fact, Drs. Dale Gerding and Lance Peterson undertook the first ever antibiotic cycling program using amikacin and gentamicin to demonstrate that withdrawal of an antibiotic to which resistance had developed would restore the activity of that drug. Humanity now faces a healthcare setting where as many as 70% of the bacterial infections afflicting patients are resistant to at least one antimicrobial that was initially active against historical bacterial ancestors. In a sense, the investigators have been preparing for this funding announcement for nearly an entire career - and are confident that the investigators can 'answer' the challenge of reversing antibacterial resistance and reducing that threat for healthcare-associated infections (HAIs). The objectives are in the main area that describes the focus for this application, which is Antimicrobial Stewardship: Preventing the development and spread of resistant organisms in the healthcare setting.

There are two specific aims for this research program to accomplish. They are:

1. Specific Aim 1: Complete development of the personalized weighted-incidence, syndromic, combination antibiogram (WISCA) tool and validate its performance as a comprehensive strategy to improve the treatment of infectious diseases for all hospitalized patients.

   - The investigators will demonstrate and expand the use of information technology based on the WISCA for the widespread use of automated clinician prompts enhancing empiric antibiotic therapy as part of a comprehensive infection control stewardship program that reduces antibiotic resistance.
2. Specific Aim 2: Demonstrate that use of such a tool improves patient outcome, lowers antimicrobial resistance and reduces cost.

   * The clinical and economic outcome measures will include changes in length of stay, duration of treatment, use of therapeutic drug monitoring, inpatient mortality, adverse events from antibacterial therapy, admission and discharge location (with the goal being fewer persons needing skilled care after discharge than is now required), 30 day readmission rates, unintended consequences from antimicrobial agent use, such as Clostridium difficile infection, antimicrobial drug cost and antimicrobial susceptibility.

All the investigator faculty are well aware of current developments in the relevant fields and are actively involved in cutting edge research that will be applied in a comprehensive, integrated fashion to solve the problem of antimicrobial resistant HAIs. The investigators look forward to working on this Large Research Project with the Agency for Healthcare Research and Quality for the improvement in the care of United States citizens.

ELIGIBILITY:
Inclusion Criteria:

* Any person admitted to the hospital with pneumonia, cellulitis, intraabdominal infection, or urinary tract infection

Exclusion Criteria:

* Any person without the 4 studied infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9673 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in length of stay | 36 months
  Changes in length of hospital stay (in days) between intervention and control groups
Rapid response to initial therapy | 36 Months
  Duration of treatment (in days) between intervention and control groups
Reduced cost of ancillary testing | 36 months
  Rate of use of therapeutic drug monitoring between intervention and control groups - ancillary testing such as therapeutic drug monitoring adds to cost of anti-infective therapy and use of fewer antibiotics when they are not needed is expected to reduce this cost
Lower mortality | 36 months
  Rate of inpatient mortality between intervention and control groups
Reduced adverse events | 36 months
  Rate of adverse events from antibacterial therapy between intervention and control groups
Improved response to Infectious Disease therapy | 36 months
  Rate of change between admission and discharge location (with the goal being fewer persons needing skilled care after discharge than is now required) between intervention and control groups - improved therapy is expected to give a better response and permit patients to return home rather than needing to go to a skilled nursing facility following their inpatient therapy
Reduced occurrence of infection recurrence | 36 months (the total time frame of the crossover study)
  30 day readmission rates (for repeated infection therapy) between intervention and control groups is a measure that is expected to differentiate between patients who receive optimal therapy that avoids recurrence of infection from those who do not
Fewer unintended consequences of antibiotic use | 36 months
  Rates of Clostridium difficile infection between intervention and control groups - antibiotic use is the main cause of the unintended consequence of Clostridium difficile infection and less antibiotic use is expected to have a lower rate of Clostridium difficile infection in the intervention group
Reduced therapy cost | 36 months
  Antimicrobial drug cost between intervention and control groups
Less antimicrobial resistance | 36 months
  Antimicrobial resistance rates between intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Lance R Peterson, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem Research Institute, Evanston, Illinois, United States